CLINICAL TRIAL: NCT03166839
Title: Management of Postpartum Haemorrhage and Effect of Geographic Region: A Secondary Analysis of the World Maternal Antifibrinolytic (WOMAN) Trial
Brief Title: Management of Postpartum Haemorrhage and Effect of Geographic Region
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 12049
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Postpartum Hemorrhage
Keywords: maternal health; statistical analysis plan
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Region 1: Africa: Women living in and experiencing PPH in countries located in Africa.
  Interventions: Other: Experiencing PPH
- Region 2: Asia: Women living in and experiencing PPH in countries located in Africa.
  Interventions: Other: Experiencing PPH
- Region 3: Europe, NA, SA, Aus: Women living in and experiencing PPH in countries located in Africa.
  Interventions: Other: Experiencing PPH

INTERVENTIONS:
Other: Experiencing PPH — No intervention given

SUMMARY:
Background: Maternal deaths occur universally and are largely avoidable. Postpartum haemorrhage accounts for a disproportionate amount of maternal deaths. There remains a great need to expeditiously decrease the rate of postpartum haemorrhage to prevent further mortality.

Methods: This study is a cohort analysis of data collected for the pragmatic international multi-centre randomized double blind placebo controlled design WOMAN Trial. It will present a univariate analysis of patient and delivery characteristics (age, type of delivery, placenta fully delivered, primary cause of haemorrhage, severity of haemorrhage), physiologic characteristics (systolic blood pressure, estimated blood loss, clinical signs of haemodynamic instability) and management characteristics (receipt of blood products, uterotonics). Multivariable logistic regression models and likelihood ratio tests will be used to examine the evidence for interaction between death from PPH and region after adjusting for any independent effects of 1) systolic blood pressure 2)age 3) type of delivery 4) receipt of blood products Discussion: This analysis of the WOMAN trial dataset will explore the relationship between geographical location, patient and environment characteristics and outcomes of postpartum haemorrhage. A protocol and statistical analysis plan is presented here.

DETAILED DESCRIPTION:
Global burden of disease Maternal deaths occur universally and are largely avoidable(1). According to the first publication of the Maternal Health Series published in the Lancet October 2016, approximately 300,000 maternal deaths occurred in the past year. Postpartum haemorrhage was the cause of one tenth of these deaths(2,3). While this number has decreased globally since 1990, haemorrhage still accounts for a disproportionate amount of maternal deaths. There remains a great need to expeditiously decrease the rate of postpartum haemorrhage to prevent further mortality.

Why study postpartum haemorrhage? The most severe outcome of postpartum haemorrhage (PPH) is the death of a mother. The World Health Organization defines maternal death as "death of a woman while pregnant or within 42 days of termination of pregnancy" (4). The clinical definition of postpartum haemorrhage refers to more than 500mL of blood loss after a vaginal delivery and more than 1000mL after a caesarean section(5). Haemorrhage is a rapidly fatal condition, most commonly caused by uterine atony, or the inability of the uterus to contract, constricting the network of vessels in the uterine muscle, gradually slowing active bleeding. For this reason, research efforts have been directed at minimizing or preventing uterine atony through preventative or treatment measures targeted at the third stage of labour(6,7). Anti-fibrinolytics have been proposed as an alternative method of slowing bleeding and have been studied both as a prophylactic intervention and a treatment modality(8-11). Risk of death from postpartum haemorrhage increases if the woman is anaemic as she cannot tolerate blood loss to the same extent that her counterparts with normal haemoglobin levels can(3,12). Recent publication of preliminary findings of the woman trial suggest that the anti-fibrinolytic tranexamic acid may reduce maternal mortality from PPH by over one third(13).

Why stratify by region? While the absolute number of maternal deaths around the world is impressive, quoting a global rate does not accurately reflect the burden of illness in different regions of the world. In developed countries like the United States of America, the risk of dying from postpartum haemorrhage after delivering a live baby is 13.4% (pooled, range: 4.7-34.6). This stands in stark contrast to the African experience, where studies have documented maternal death rates from PPH to be as high as 33.9% (pooled, range: 13.3-43.5)(14). There are other reasons why these numbers can vary so broadly. An obvious hypothesis is that more women die from postpartum haemorrhage in developing countries than their counterparts in developed countries because it is more prevalent, more severe or is managed differently than in other parts of the world. It has been proposed, however, that the different rates in fact reflect a paucity of reliable data that is region specific. This is indeed the case when we look at the continent of Africa, where studies done to date capture only the experiences of eight of the 54 countries on the continent (Egypt in the North, Senegal in the West, and the Democratic Republic of Congo, South Africa, Tanzania, Zambia, Zimbabwe in the East and South)(14). A third factor in estimating deaths from postpartum haemorrhage reflects the different birthing environments across regions. In some countries, up to 50% of women deliver at home with support from a traditional birth attendant and never access a medical clinic or hospital. When most women do not deliver in a hospital or clinic, they do not die in a hospital or clinic so their data goes largely unregistered(9). Despite the fact that the "poorest countries have the poorest data"(12) enough is known about postpartum haemorrhage to inform action and spur further investigation, as many organizations have done(15).

While developing countries carry a higher burden of maternal deaths from postpartum haemorrhage, the impact of maternal death from PPH does not spare the developed world(14). Haemorrhage remains a leading cause of maternal death in countries where the majority of deliveries are performed in hospital with highly skilled support(16). This may be, in part, due to the unpredictability of postpartum haemorrhage, even in low-risk women(12). Risk factors for postpartum haemorrhage are commonly accepted to include previous postpartum haemorrhage, pre-eclampsia, disorders of the placenta, induction or augmentation of labour, perineal trauma, high birthweight and retained products(7)(16). Further, reporting occurrence of postpartum haemorrhage varies due to varying definitions of blood loss, the way blood loss is measured, intra-partum management strategies including uterotonics, uterine massage, and cord traction, interventions including method of delivery as well as the underlying characteristics of the population being studied(6)(3). Much time and resources have been invested in investigating the use of uretonics such as oxytocin to treat the most common causes of postpartum haemorrhage(7).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16 years and older
* Clinical diagnosis of postpartum haemorrhage (PPH) after vaginal delivery or caesarean section
* "clinical uncertainty" about benefit of tranexamic acid in addition to routine management of PPH

Exclusion Criteria:

- Women aged 16 years and older with a clinical diagnosis of postpartum haemorrhage with clear indication or contra-indication for tranexamic acid

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Eligible adult women with a clinical diagnosis of postpartum haemorrhage following vaginal or caesarean section delivery will be included in this cohort analysis. While the diagnosis was clinical, a definition of postpartum haemorrhage could be based on clinically estimated blood loss of more than 500mL after vaginal birth or 1000mL after caesarean section or any blood loss sufficient to compromise haemodynamic stability.
Sampling Method: Probability Sample
Enrollment: 20060 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Death | Within 42 days of delivery
  Death due to bleeding from PPH

CONTACTS AND LOCATIONS:
Overall Officials: Ian Roberts, Principal Investigator — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham W, Woodd S, Byass P, Filippi V, Gon G, Virgo S, Chou D, Hounton S, Lozano R, Pattinson R, Singh S. Diversity and divergence: the dynamic burden of poor maternal health. Lancet. 2016 Oct 29;388(10056):2164-2175. doi: 10.1016/S0140-6736(16)31533-1. Epub 2016 Sep 16. PMID 27642022
- [Background] Calvert C, Thomas SL, Ronsmans C, Wagner KS, Adler AJ, Filippi V. Identifying regional variation in the prevalence of postpartum haemorrhage: a systematic review and meta-analysis. PLoS One. 2012;7(7):e41114. doi: 10.1371/journal.pone.0041114. Epub 2012 Jul 23. PMID 22844432
- [Background] Carroli G, Cuesta C, Abalos E, Gulmezoglu AM. Epidemiology of postpartum haemorrhage: a systematic review. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. PMID 18819848
- [Background] Begley CM, Gyte GM, Devane D, McGuire W, Weeks A. Active versus expectant management for women in the third stage of labour. Cochrane Database Syst Rev. 2015 Mar 2;(3):CD007412. doi: 10.1002/14651858.CD007412.pub4. PMID 25730178
- [Background] Mousa HA, Blum J, Abou El Senoun G, Shakur H, Alfirevic Z. Treatment for primary postpartum haemorrhage. Cochrane Database Syst Rev. 2014 Feb 13;2014(2):CD003249. doi: 10.1002/14651858.CD003249.pub3. PMID 24523225
- [Background] Shakur H, Roberts I, Edwards P, Elbourne D, Alfirevic Z, Ronsmans C. The effect of tranexamic acid on the risk of death and hysterectomy in women with post-partum haemorrhage: statistical analysis plan for the WOMAN trial. Trials. 2016 May 17;17(1):249. doi: 10.1186/s13063-016-1332-2. PMID 27188698
- [Background] McClure EM, Jones B, Rouse DJ, Griffin JB, Kamath-Rayne BD, Downs A, Goldenberg RL. Tranexamic acid to reduce postpartum hemorrhage: A MANDATE systematic review and analyses of impact on maternal mortality. Am J Perinatol. 2015 Apr;32(5):469-74. doi: 10.1055/s-0034-1390347. Epub 2014 Oct 7. PMID 25289705
- [Background] Gohel, M Efficacy of tranexemic acid in decreasing blood loss during and after cesarean section: A randomised case controlled prospective study. J Obstet Gynecol India. 2007;57(3):227-30.
- [Background] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Background] Mousa HA, Cording V, Alfirevic Z. Risk factors and interventions associated with major primary postpartum hemorrhage unresponsive to first-line conventional therapy. Acta Obstet Gynecol Scand. 2008;87(6):652-61. doi: 10.1080/00016340802087660. PMID 18568465
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Ronsmans C, Graham WJ; Lancet Maternal Survival Series steering group. Maternal mortality: who, when, where, and why. Lancet. 2006 Sep 30;368(9542):1189-200. doi: 10.1016/S0140-6736(06)69380-X. PMID 17011946
- [Result] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509